CLINICAL TRIAL: NCT05782426
Title: Efficacy and Safety of Paclitaxel Polymeric Micelles for Injection, Platinum (Cisplatin/Carboplatin) Combined With Sindilizumab Injection in the First-line Treatment of Advanced Non-squamous Non-small Cell Lung Cancer
Brief Title: Study of Polymeric Micellar Paclitaxel, Platinum Combined With Sindilizumab Injection for Advanced Non-squamous NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu Cancer Institute & Hospital (Other)
Responsible Party: Principal Investigator, Rong Yin, MD PhD, Professor, Jiangsu Cancer Institute & Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YZ-006
Record Dates: First submitted 2023-02-27; First posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Non-squamous NSCLC
Keywords: NSCLC; paclitaxel polymeric micelles for injection; sindilizumab injection
MeSH Terms: interventions — Injections; Platinum

STUDY DESIGN:
Intervention Model Description: Patients will be treated with paclitaxel polymeric micelles for injection, platinum (cisplatin/carboplatin) in combination with sindilizumab for 4-6 cycles. If patient assessment is of clinical benefit, maintenance therapy with sindilizumab plus paclitaxel polymeric micelles for injection(≤230mg/m^2) can be continued based on investor's evaluation and patient's own choice until disease progression (PD), unacceptable toxicity, withdrawal of consent, initiation of additional antineoplastic therapy, death, or other protocol-specified conditions for discontinuation of treatment, whichever comes first.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- paclitaxel polymeric micelles for injection, platinum combined with sindilizumab injection (Experimental): Patients will be treated with paclitaxel polymeric micelles for injection, platinum (cisplatin/carboplatin) in combination with sindilizumab for 4-6 cycles. If patient assessment is of clinical benefit, maintenance therapy with sindilizumab plus paclitaxel polymeric micelles for injection(≤230mg/m^2) can be continued based on investor's evaluation and patient's own choice until disease progression (PD), unacceptable toxicity, withdrawal of consent, initiation of additional antineoplastic therapy, death, or other protocol-specified conditions for discontinuation of treatment, whichever comes first.
  Interventions: Drug: paclitaxel polymeric micelles for injection

INTERVENTIONS:
Drug: paclitaxel polymeric micelles for injection — Patients will be treated with paclitaxel polymeric micelles for injection, platinum (cisplatin/carboplatin) in combination with sindilizumab for 4-6 cycles. If patient assessment is of clinical benefit, maintenance therapy with sindilizumab plus paclitaxel polymeric micelles for injection(≤230mg/m^2) can be continued based on investor's evaluation and patient's own choice until disease progression (PD), unacceptable toxicity, withdrawal of consent, initiation of additional antineoplastic therapy, death, or other protocol-specified conditions for discontinuation of treatment, whichever comes first.
  Other Names: platinum; sindilizumab injection

SUMMARY:
This is a prospective, single-arm, single-center, phaseⅡtrial to evaluate the efficacy and safety of Paclitaxel Polymeric Micelles for Injection, platinum (cisplatin/carboplatin) in combination with sindilizumab injection as first-line chemotherapy in advanced or metastatic non-squamous NSCLC patients without EGFR mutation or ALK rearrangement.

DETAILED DESCRIPTION:
Patients with histologically or cytologically confirmed metastatic or recurrent stage ⅢB/Ⅳ non-squamous NSCLC, inoperable or inappropriate for radical concurrent chemoradiotherapy, and without previous systemic treatment will be screened after signing Informed Consent. Patients will be treated with paclitaxel polymeric micelles for injection, platinum (cisplatin/carboplatin) in combination with sindilizumab for 4-6 cycles. If patient assessment is of clinical benefit, maintenance therapy with sindilizumab plus paclitaxel polymeric micelles for injection (≤230mg/m^2) can be continued based on investor's evaluation and patient's own choice until disease progression (PD), unacceptable toxicity, withdrawal of consent, initiation of additional antineoplastic therapy, death, or other protocol-specified conditions for discontinuation of treatment, whichever comes first.

Patients receiving sindilizumab who has first radiologic evidence of PD according to RECIST 1.1 can continue the treatment if their clinical status is stable, without evidence of rapid radiologic progression and if they are deemed by the investigator to be continuing to benefit from the treatment. Re-evaluation by imaging is required after a minimum interval of 4 weeks (±7 days), if PD is confirmed by the re-evaluation, the study treatment should be stopped. If PD is not confirmed, the study treatment can be continued, with assessments at the planned time points for imaging as specified in the protocol, until PD is confirmed on imaging.

The maximum treatment duration of sindilizumab injection and paclitaxel polymeric micelles for injection is 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be signed before implementing any trial-related procedures;
2. Age ≥18 years old;
3. Patients with histologically or cytologically confirmed metastatic or recurrent (stage IIIB/IV) non-squamous NSCLC (International Association for the Study of Lung Cancer and American Joint Committee on Classification of Cancer, 8th Edition TNM staging), inoperable or inappropriate for radical concurrent chemoradiotherapy, and without previous systemic treatment；
4. No EGFR gene sensitive mutation or ALK gene fusion mutation is confirmed by histological specimens; PD-L1 immunohistochemical results is required before enrollment; There is no special restriction on the source of genetic test report.
5. According to the Response Evaluation Criteria in Solid Tumors (RECIST, version 1.1), there is at least one radiographically measurable lesion. Lesions located in the area of previous radiotherapy can be considered as measurable lesions if the progression is confirmed.
6. Have not received any previous systemic antitumor therapy for advanced/metastatic diseases. Participants who have previously received platinum-based adjuvant/neoadjuvant chemotherapy, or radical chemoradiotherapy for advanced disease are allowed to enroll if the interval between disease progression or recurrence and the end of the last chemotherapy treatment is at least 6 months.
7. Patients are allowed to receive palliative radiotherapy provided that it is completed 7 days before the first study treatment and the radiotherapy-related toxicity have recovered to grade 1 or less (CTCAE5.0);
8. ECOG score: 0-1
9. Expected survival time > 3 months
10. Normal organ function, patients should meet the following laboratory indicators:

1)Blood routine test should meet the following criteria (no blood transfusion, no use of blood products, granulocyte colony-stimulating factor, or other hematopoietic growth factors within 7 days before blood routine test); White blood cell count ≥3.0x10^9/L, absolute neutrophil count (ANC) ≥1.5x10^9/L，Platelet count ≥100×10^9/L，Hemoglobin >9g/dL. If patients receive blood component transfusion (red blood cells, platelets, etc.) during the screening period, blood routine test should be performed again at an interval of 1 week to meet the above criteria before continuing screening.

2) Blood biochemical examination must meet the following criteria: Total bilirubin ≤1.5 times the upper limit of normal (ULN), and aspartate aminotransferase (AST), alanine aminotransferase (ALT), or alkaline phosphatase (ALP) ≤2.5 times ULN (ALT, AST, or ALP≤ 5×ULN for patients with liver metastases, and ALP≤10×ULN for patients with bone metastases); Serum creatinine ≤1.5 times ULN and creatinine clearance (calculated using Cockcroft-Gault formula) ≥60 ml/min； 3) Normal coagulation function, defined as international normalized ratio (INR) or prothrombin time (PT) ≤1.5 times ULN; 4) Normal thyroid function, defined as thyroid stimulating hormone (TSH) within the normal range. Subjects with baseline TSH beyond the normal range, but total T3 (or FT3) and FT4 are within the normal range can also be enrolled; 5) Myocardial zymogram within the normal range (if the investor judges that the simple laboratory result is not of clinical significance, the patient is allowed to be included); 11.For female patients of childbearing age, a negative urine or serum pregnancy test should be performed within 3 days before the first study drug administration (day 1 of cycle 1). If the urine pregnancy test result cannot be confirmed as negative, a blood pregnancy test is requested. Female patients who are not of childbearing age are defined as those who have been postmenopausal for at least 1 year or have undergone surgical sterilization or hysterectomy; 12.If there is a risk of conception, all patients (male or female) are required to use contraception throughout the treatment period until 180 days after the last study drug administration.

Exclusion Criteria:

1. Patients with small cell lung cancer (SCLC, including SCLC mixed with NSCLC), squamous non-small cell lung cancer; Non-squamous NSCLC with EGFR gene sensitive mutation and ALK gene fusion mutation;
2. Patients who have received radiation therapy before the first administration of study drug, and if one of the following conditions occurred:

1) ≥30% of bone marrow have received radiotherapy within 14 days prior to treatment; 2) Radiation to a lung lesion at a dose of >30Gy within 6 weeks before treatment( to be eligible, patients must have recovered to grade 1 or lower from previous radiation toxicity, no need for glucocorticoids, and no history of radiation pneumonitis); 3)Palliative radiation therapy completed within 7 days before the first study drug administration.

3.Malignant diseases other than NSCLC diagnosed within 5 years before the first dose (excluding radical basal cell carcinoma, squamous carcinoma, and/or radical resection carcinoma in situ); 4.Currently participating in an interventional clinical study treatment, or receiving other study drugs or using study devices within 4 weeks before the first dose； 5.Previous treatment with anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or agent targeting another stimulatory or synergistic T-cell receptor (e.g., CTLA-4, OX-40, CD137)； 6.Received systemic treatment with Chinese drugs or immunomodulatory drugs (including thymosin, interferon and interleukin, except for local use to control pleural effusion) with anti-NSCLC indications within 2 weeks before the first dose; 7.An active autoimmune disease requiring systemic therapy (e.g., disease-modifying agents, glucocorticoids, or immunosuppressants) occurred within 2 years before the first dose. Alternative therapies (e.g., thyroxine, insulin, or physiological glucocorticoids for adrenal or pituitary insufficiency) is not considered systemic therapy; 8.Receiving systemic glucocorticoid therapies (excluding topical glucocorticoids by nasal spray, inhalation, or other route)) or any other form of immunosuppressive therapies within 7 days before the first medication of the study; Note: Physiological doses of glucocorticoids (≤10 mg prednisone/day or equivalent) are permitted； 9.Patients with active or untreated central nervous system (CNS) metastasis;

1. If the patient's CNS tumor metastasis is confined to supratentorial and/or cerebellum, has been adequately treated, and has been clinically stable (imaging testing, enhanced MRI or CT is preferred) for at least 4 weeks, Participants are eligible for the study if they have recovered to NCI-CTC AE ≤ grade1 at least 2 weeks before the first dose of medication. If new asymptomatic CNS metastases are detected on screening scans, radiation therapy and/or surgery for CNS metastases are required;
2. Glucocorticoid therapy is not required, or glucocorticoid therapy is discontinued within 7 days before the first dose, or glucocorticoid dosage is stable and reduced to less than 10mg prednisone per day (or equivalent) within 7 days before the first dose.

10.Spinal cord compression without radical treatment with surgery and/or radiotherapy, or previously diagnosed spinal cord compression without clinical evidence of stable disease for ≥4 weeks before enrollment; 11.Patients with clinically uncontrollable pleural effusion/peritoneal effusion (patients who did not need to drain effusion or stopped drainage for 3 days without significant increase in effusion could be enrolled); 12.Known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation; 13.Patients with known allergies to sindilizumab, paclitaxel polymeric micelles for injection, platinum (cisplatin/carboplatin) and other active ingredients or excipients; 14.Patients who have not fully recovered from any intervention-related toxicity and/or complications before starting treatment (i.e., grade ≤1 or baseline, excluding fatigue or alopecia); 15.Patient with a history of human immunodeficiency virus (HIV) infection (i.e., HIV 1/2 antibody positive); 16.Patient who has untreated active hepatitis B (defined as both HBsAg positivity and HBV-DNA copies greater than the upper limit of normal range in the laboratory of the participating center);

Note: Patient with hepatitis B who meets the following criteria are also eligible for inclusion:

1. Patients with HBV viral load <1000 copies /ml (200 IU/ml) before the first study medication should receive anti-HBV therapy throughout the study chemotherapy to avoid viral reactivation;
2. For patients with anti-HBc (+), HBsAg (-), anti-hbs (-) and HBV viral load (-), prophylactic anti-HBV therapy is not required, but viral reactivation should be closely monitored.

17.Active HCV-infected patients (positive for HCV antibodies and HCV-RNA levels above the upper limit of detection); 18.Patients who have received a live vaccine within 30 days before the first dose of study drug (cycle 1, day 1); Note: Administration of injectable inactivated virus vaccine against seasonal influenza within 30 days before the first dose of study is allowed; Live, attenuated, intranasal influenza vaccine is not allowed.

19.Pregnant or lactating women; 20.The presence of any serious or uncontrolled systemic illness, such as:

1）significant rhythm, conduction or morphological abnormalities in resting ECG, such as complete left bundle branch block, ≥II degree heart block, ventricular arrhythmia or atrial fibrillation; 2）Unstable angina, congestive heart failure, New York Heart Association (NYHA) grade ≥ 2 chronic heart failure; 3）Myocardial infarction within 6 months before enrollment; 4）Poor blood pressure control (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg)； 5）Patient with a history of noninfectious pneumonia requiring glucocorticoid treatment within 1 year before the first dose, or current clinically active interstitial lung disease; 6）Active pulmonary tuberculosis; 7）Presence of active or uncontrolled infection requiring systemic therapy; 8）Presence of clinically active diverticulitis, abdominal abscess, and gastrointestinal obstruction; 9）Presence of liver diseases such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis; 10）Poorly controlled diabetes (fasting blood glucose (FBG) > 10mmol/L); 11）Patient whose urine routine test shows urinary protein ≥++ and confirmed 24-hour urinary protein quantitation > 1.0 g; 12）Patients with a mental disorder who is unable to cooperate with treatment; 21.Patients who have medical history or evidence of disease, treatment or laboratory abnormalities, or other conditions deemed by the investigator to be inappropriate for enrollment that may interfere with the results of the trial or preclude full participation in the study.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-03-15 (Estimated); Primary Completion 2024-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the Objective Response Rate (ORR) | From the first dose of study drug to the first date of documentation of disease progression or death whichever occurred first ,up to approximately 2 years
  Objective Response Rate (ORR) Based on RECIST 1.1 assessed by investigator review, the proportion (%) of patients with confirmed best overall response of complete response (CR) or partial response (PR)

SECONDARY OUTCOMES:
To evaluate the Disease Control Rate (DCR) | From the first dose of study drug to the first date of documentation of disease progression or death whichever occurred first,up to approximately 2 years
  Disease Control Rate (DCR) Based on RECIST 1.1 assessed by investigate review ,the proportion (%) of patients with at least one visit response of complete response (CR) or partial response (PR), or stable disease (SD).
To evaluate the Duration of Response (DOR) | From date of first documented confirmed CR or PR until date of first documentation of PD or death whichever occurred first, up to approximately 2 years
  Duration of Response (DOR) was defined as the time from the first documentation of CR or PR to the date of first documentation of PD or death (whichever occurred first) in participants with confirmed CR or PR based on RECIST 1.1 assessed by investigator review.
To evaluate the Progression-free Survival (PFS) | From the first study dose date to the date of first documentation of disease progression or death (whichever occurred first), up to approximately 2 years
  Progression-free Survival (PFS) was defined as the time from the first study dose date to the date of first documentation of disease progression or death (whichever occurred first) based on RECIST 1.1 assessed by investigator review. PD was defined as at least a 20% increase in the sum of LD of target and non-target lesions as compared with the smallest sum of LD and the increase of LD was at least 5 mm (including new lesions).
To evaluate the Overall Survival (OS) | From the date of first dose of study drug until date of death from any cause (up to approximately 5 years )
  Overall Survival (OS) was measured from the date of first dose of study drug until date of death from any cause. Participants who were lost to follow-up and the participants who were alive at the date of data cutoff was censored at the date the participant was last known alive, whichever came earlier.
To evaluate the Safety | From first dose until 30 days after the last dose, up to approximately 2 years
  Safety was measured by number and grade of adverse events Number of Participants With adverse events (AE), Treatment-releated Adverse Events (TRAEs) , Serious Adverse Events (SAEs) and immune-related adverse events (irAE) , events will be classified according to CTCAE V5.0

CONTACTS AND LOCATIONS:
Overall Officials: Jifeng Feng, Study Chair — Affiliated to Jiangsu Cancer Hospital & Institute
Locations (2):
- China (2):
  - Jiangsu Cancer Institute & Hospital, Nanjing, Jiangsu
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No